CLINICAL TRIAL: NCT00814775
Title: Comparison Between the Fastrach and CTrach Laryngeal Mask Airway for Intubation of Patients With a Mallampati Score 3 or 4
Brief Title: Comparison Between the Fastrach and CTrach Laryngeal Mask Airway
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment challenges, device no longer available
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 08-358
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Intubation
Keywords: Laryngeal mask; Difficult intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Fastrach Laryngeal Mask Airway intubation
  Interventions: Device: Fastrach Laryngeal Mask
- Group 2 (Active Comparator): Intubation of difficult airway using CTrach Laryngeal Mask
  Interventions: Device: CTrach Laryngeal Mask

INTERVENTIONS:
Device: Fastrach Laryngeal Mask — Intubation of difficult airway using Fastrach Laryngeal Mask
  Arms: Group 1
Device: CTrach Laryngeal Mask — CTrach Laryngeal Mask intubation
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine the effectiveness of the Fastrach and the CTrach Laryngeal mask airway to achieve placement of a breathing tube in the windpipe of patients where this may be difficult.

DETAILED DESCRIPTION:
Participant will be randomly assigned to receive one of 2 conventional airway devices - the Fastrach Laryngeal Mask Airway or the CTrach Laryngeal Mask Airway. This study will compare the time required for successful intubation between the two devices.

Postoperative visit will be performed to assess the participant's clinical condition and to receive participant's feed back.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an ASA score of 1-3.
2. Scheduled for elective surgical procedure
3. Age 18 and above
4. Patients with Mallampati airway classification scores III and IV

Exclusion Criteria:

1. Current pregnancy
2. Patients undergoing brain aneurysm clipping brain arteriovenous malformation surgery or vascular surgery procedures
3. Patients with obstructive sleep apnea or with a history of difficult ventilation
4. Mouth opening less than 3 cm.
5. Patients with indication for awake fiberoptic intubation or with a history of difficult intubation
6. Patients with cancer of the neck or the upper airway
7. Emergent surgery, patients requiring rapid sequence induction
8. Patients with severe gastroesophageal reflux
9. Patients with severe cardiac, pulmonary, hepatic or renal co-morbidities. 10. Patients unable to consent their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maurtua, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fastrach: Fastrach Laryngeal Mask Airway intubation
  Fastrach Laryngeal Mask: Intubation of difficult airway using Fastrach Laryngeal Mask
- CTrach: Intubation of difficult airway using CTrach Laryngeal Mask
  CTrach Laryngeal Mask: CTrach Laryngeal Mask intubation
Period: Overall Study
Arm/Group | Fastrach | CTrach
Started | 23 | 20
Completed | 23 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fastrach | CTrach | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (16) | 59 (15) | 59 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Time Required for Successful Intubation Between the Fastrach and CTrach LMA Devices in Patients With a Mallampati Score III and IV Without Use of Fiberoptic Bronchoscopy
Time Frame: from start of intubation to successfully intubated
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Fastrach | CTrach
Number analyzed (Participants) | 23 | 20
seconds | 41 [31 to 78] | 40 [32 to 55]
Statistical Analysis 1: Comparison: Fastrach vs CTrach; Test type: Superiority or Other; p = 0.72, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.55 to 2.37] — CTrach vs. Fastrach

2. Primary Outcome: To Compare the Time Required for Successful Intubation Between the Fastrach and CTrach LMA Devices in Patients With a Mallampati Score III and IV Use of Fiberoptic Bronchoscopy
Time Frame: 60 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Fastrach | CTrach
Number analyzed (Participants) | 23 | 20
seconds | 35 [28 to 43] | 40 [32 to 51]
Statistical Analysis 1: Comparison: Fastrach vs CTrach; Test type: Superiority or Other; p = 0.45, Regression, Cox; Cox Proportional Hazard = 0.76, 95% CI 2-sided [0.38 to 1.54] — CTrach vs. Fastrach

ADVERSE EVENTS:
Arm/Group | Fastrach | CTrach
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No